CLINICAL TRIAL: NCT01007916
Title: Subjective Evaluation of a Commercially Marketed Contact Lens Amongst a Subset of the Contact Lens Wearing Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-336-C-016
Record Dates: First submitted 2009-11-02; First posted 2009-11-05 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon B / Habitual (Other): Lotrafilcon B contact lenses worn first, with habitual contact lenses worn second. Both products worn bilaterally as often as is typical for habitual lenses, and in the same modality as is typical for habitual lenses, as prescribed by regular eye care practitioner, with extended wear not to exceed 6 nights.
  Interventions: Device: Lotrafilcon B contact lens; Device: Habitual contact lens
- Habitual / Lotrafilcon B (Other): Habitual contact lenses worn first, with lotrafilcon B lenses worn second. Both products worn bilaterally as often as is typical for habitual lenses, and in the same modality as is typical for habitual lenses, as prescribed by regular eye care practitioner, with extended wear not to exceed 6 nights.
  Interventions: Device: Lotrafilcon B contact lens; Device: Habitual contact lens

INTERVENTIONS:
Device: Lotrafilcon B contact lens — Commercially marketed, silicone hydrogel, spherical contact lens having a recommended replacement schedule of monthly.
Device: Habitual contact lens — Habitual soft spherical contact lens having a recommended replacement schedule of 2 weeks or monthly.

SUMMARY:
The purpose of this study is to compare the performance of commercially marketed contact lenses to habitual contact lenses in a selected segment of the contact lens wearing population.

ELIGIBILITY:
Inclusion Criteria:

* Habitual spherical soft contact lens wearer who wears a contact lens with a recommended replacement schedule of 2 weeks or monthly.
* Wears lenses at least 5 days per week and at least 12 hours per day.
* Removes contact lenses daily or, if prescribed by their regular eye care practitioner, sleeps overnight in contact lenses no more than 6 consecutive nights.
* Reports 2 or fewer common lens-related symptoms with current contact lenses with a frequency of "frequently" or "always".
* Able to achieve distance visual acuity of at least 20/40 in each eye at the dispense of each pair of study lenses.
* Has acceptable or optimal fit for each eye at the dispense of each pair of study lenses.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Currently sleeping in contact lenses for more than 6 consecutive nights.
* Currently wearing daily disposable contact lenses and certain protocol-specified lens brands.
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled but not dispensed due to failing inclusion/exclusion criteria. This participant is included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Period: Period 1, 4 Weeks of Wear
Arm/Group | Lotrafilcon B / Habitual | Habitual / Lotrafilcon B
Started | 23 | 26
Completed | 22 | 26
Not Completed | 1 | 0
Not completed — Failed inclusion/exclusion | 1 | 0
Period: Period 2, 4 Weeks of Wear
Arm/Group | Lotrafilcon B / Habitual | Habitual / Lotrafilcon B
Started | 22 | 25 (One participant completed Period 1 but did not start Period 2 due to failing inclusion criteria.)
Completed | 21 | 25
Not Completed | 1 | 0
Not completed — Relocation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This reporting group includes all enrolled and dispensed subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 30.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Comfort Upon Insertion
Description: Comfort upon insertion, as interpreted by the participant, was recorded on a questionnaire by the participant using a 10-point scale, with 1 being poor and 10 being excellent. Comfort upon insertion was assessed as a single, retrospective evaluation of 4-weeks' wear time.
Time Frame: 4 weeks of wear
Population: Analysis conducted per protocol, with exclusions due to major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Lotrafilcon B: Commercially marketed, silicone hydrogel, spherical contact lens having a recommended replacement schedule of 30 days.
- Habitual: Habitual soft spherical contact lens having a recommended replacement schedule of 2 weeks or monthly.
Arm/Group | Lotrafilcon B | Habitual
Number analyzed (Participants) | 47 | 46
Units on a Scale | 8.7 (2.0) | 9.2 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 86 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Lotrafilcon B | Habitual
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48

LIMITATIONS AND CAVEATS:
Participants were masked to lotrafilcon B lenses only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.